CLINICAL TRIAL: NCT06934395
Title: Sustaining Healthy Choices: Optimizing a State-wide Scalable Intervention to Improve Alcohol and HIV Self-management in Adolescents and Emerging Adults
Brief Title: SHARE Program: SUSTAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: University of Florida (Other); Northeastern University (Other); University of Michigan (Other); University of South Florida (Other); CAN Community Health (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sylvie Naar, Principal Investigator, Florida State University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002536; 5P01AA029547 (NIH)
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Within-participant micro-randomization - Prompt (Experimental): Participants will be randomized daily to receive a text messaged prompt focused on medication adherence or stress.
  Interventions: Behavioral: Text Message Prompts
- Within-participant micro-randomization - No Prompt (No Intervention): Participants will be randomized daily to not receive a text messaged prompt focused on medication adherence or stress.
- Between-participant randomization - CIAS + Week 2 Coaching Session (Experimental): Participants will be randomized at the end of week 2 (day 14) to receive the Healthy Choices telehealth intervention with trained interventionist at week 2.
  All enrolled participants will receive an initial Healthy Choices mHealth intervention which involves a MI based coaching session via Computerized Intervention Authoring Software (CIAS).
  Interventions: Behavioral: Healthy Choices
- Between-participant randomization - CIAS + No Week 2 Coaching Session (No Intervention): Participants will be randomized at the end of week 2 (day 14) to NOT receive the Healthy Choices telehealth intervention with trained interventionist at week 2.
  All enrolled participants will receive an initial Healthy Choices mHealth intervention which involves a MI based coaching session via Computerized Intervention Authoring Software (CIAS).

INTERVENTIONS:
Behavioral: Healthy Choices — Healthy Choices is an adapted and developmentally tailored intervention designed to address self-management of risk behaviors and HIV from Motivational Enhancement Therapy, a brief alcohol intervention in SAMHSA's registry of evidenced-based programs. For the purposes of this project, this intervention will be delivered as a combination approach, with all participants receiving an initial session via CIAS, and randomized to either receiving a telehealth session with a trained interventionist at week 2, with additional randomizations for telehealth sessions at weeks 4 and 6. The goal is to test if delivering (vs. not delivering) a coaching session increases the likelihood of achieving viral suppression and meeting criteria for no risky alcohol use at month 3
  Arms: Between-participant randomization - CIAS + Week 2 Coaching Session
Behavioral: Text Message Prompts — This within-participant micro-randomization will test whether, on average, delivering (vs. not delivering) a text messaged prompt focused on medication adherence or stress increases the likelihood of medication adherence by the end of the current day .
  Arms: Within-participant micro-randomization - Prompt

SUMMARY:
The goal of PROJECT SUSTAIN is to optimize Healthy Choices to advance an adaptive and scalable intervention designed to improve self-management of alcohol and HIV in Young People with HIV (YPWH) while understanding the context for state-wide implementation and sustainment in a Hybrid Experimental Design (HED). SUSTAIN utilizes mHealth and telehealth intervention delivery of Healthy Choices (HC), combined with text messaging between sessions, to increase the likelihood of daily medication adherence (primary outcome), and increase the likelihood of achieving viral suppression and meeting criteria for no risky alcohol use at month 3 (secondary outcome).

DETAILED DESCRIPTION:
Primary aim: To test whether, on average, delivering (vs. not delivering) a text messaged prompt focused on medication adherence or stress increases the likelihood of medication adherence by the end of the current day.

Secondary aim: To test whether offering (vs. not offering) a Healthy Choices telehealth coaching session at the end of week 2 (day 14) increases the likelihood of achieving viral suppression and meeting criteria for no risky alcohol use at month 3.

Implementation Aim: Assess barriers and facilitators to the implementation and sustainment of intervention sequences for state-wide scale up using mixed methods (EPIS qualitative interviews, youth satisfaction and dose received, fidelity for telehealth, paradata for mHealth, and cost-effectiveness analysis).

Cross-project Moderator Aim: Explore age, biological sex and gender, ethnicity, other substance use, and mental health as moderators of intervention effects.

Primary hypothesis to be tested: Delivering (vs. not delivering) a text messaged prompt will lead to greater likelihood of medication adherence by the end of the current day.

Secondary hypothesis to be tested: Offering a Healthy Choices telehealth coaching at the end of week 2 will lead to greater likelihood of achieving viral suppression and meeting criteria for no risky alcohol use at month 3 (post-intervention) compared to not offering a Healthy Choices telehealth coaching session at the end of week 2.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years and 0 months to 29 years and 11 months.
* Currently reside in Florida
* History of alcohol use
* Are not pregnant nor trying to conceive within the study's timeline
* Are able to read and understand English
* Have internet access via smartphone, tablet or computer
* Are willing to provide informed consent.

Exclusion Criteria:

* Adults unable to consent
* Prisoners
* Those using long-acting injectables as HIV medication regimen

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
ART Adherence | Daily for 56 Days
  Antiretroviral (ART) adherence will be assessed daily using an Ecological Momentary Assessment (EMA) survey delivered via SMS. Individuals will be asked whether they took some or all of their medication.

SECONDARY OUTCOMES:
Alcohol Use | Baseline, 3 month, and 6 month
  Alcohol will be assessed using the Timeline Followback (TLFB) measure to capture amount of drinking over a 30 day period, assessed at baseline, and at the 3 and 6 month follow-ups. Participants complete a 30 day calendar that assesses number of drinks per day and number of hours spent drinking per drinking day.
HIV Viral Load | Baseline, 3 month, and 6 month
  HIV Viral Load collected via Dried Blood Spot (DBS) kits. The limit of detection (LOD) of the m2000 test is 832 copies/mL or Log 2.92 copies/mL. For samples with VL above the LOD (>Log 2.92) can be quantified so a VL is provided. In case of samples with less than LOD is given as <2.92 but it's reported as detected as the presence of HIV virus is detected but cannot be quantified as it's below the LOD so cannot be measured. And samples that are not detected are reported as 'not detected.'

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Florida State University, Center for Translational Behavioral Science, Tallahassee, Florida
  - University of South Florida, Tampa, Florida
  - Northeastern University, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan